CLINICAL TRIAL: NCT04584671
Title: Lung Structure-Function In SurVivors of Mild and SEvere COVID-19 Infection: 129Xe MRI and CT For Rapid Evaluations and NExt-wave Healthcare Planning
Brief Title: Lung Structure-Function In Survivors of Mild and Severe COVID-19 Infection
Acronym: LIVECOVIDFREE
Status: Active, not recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Grace Parraga, PhD, Scientist. Robarts Research Institute, Western University, Canada
Other Study IDs: ROB0050
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Covid19
Keywords: Covid19; Pulmonary Function; Xenon-129; Magnetic Resonance Imaging
MeSH Terms: conditions — COVID-19 | interventions — Tomography, X-Ray Computed; Respiratory Function Tests; Walk Test; Hematologic Tests; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mild COVID-19 Infection Group: 100 participants age ≥ 18 and <80 years who experienced a documented case (documented by positive COVID-19 test and/or clinical history) of mild COVID-19 infection, all of whom are within 3 months post recovery and non-infectious.
  Interventions: Diagnostic Test: Hyperpolarized Xenon-129 MRI of the lungs; Diagnostic Test: Computed Tomography (CT); Diagnostic Test: Pulmonary Function Tests (PFT); Diagnostic Test: Six Minute Walk Test (6MWT); Diagnostic Test: Sputum analysis; Diagnostic Test: Blood analysis; Other: Questionnaires
- Severe COVID-19 Infection Group: 100 participants age ≥ 18 and <80 years who experienced a documented case (documented by positive COVID-19 test and/or clinical history) of severe COVID-19 infection, including at least 50 participants who were hospitalized with COVID-19 infection, all of whom are within 3 months post recovery and non-infectious.
  Interventions: Diagnostic Test: Hyperpolarized Xenon-129 MRI of the lungs; Diagnostic Test: Computed Tomography (CT); Diagnostic Test: Pulmonary Function Tests (PFT); Diagnostic Test: Six Minute Walk Test (6MWT); Diagnostic Test: Sputum analysis; Diagnostic Test: Blood analysis; Other: Questionnaires

INTERVENTIONS:
Diagnostic Test: Hyperpolarized Xenon-129 MRI of the lungs — Participants will be imaged using MRI using hyperpolarized xenon-129 gas as a contrast gas
  Other Names: 129Xe MRI
Diagnostic Test: Computed Tomography (CT) — Participants will undergo a CT scan of the thoracic cavity
  Other Names: CT
Diagnostic Test: Pulmonary Function Tests (PFT) — Participants will have their lung function evaluated using PFT
  Other Names: PFT
Diagnostic Test: Six Minute Walk Test (6MWT) — Participants will perform the six minute walk test as a measure of exercise capacity
  Other Names: 6MWT
Diagnostic Test: Sputum analysis — Participants will provide a sputum sample that will be analysed for eosinophils
Diagnostic Test: Blood analysis — Participants will have their blood drawn and analysed for eosinophil count.
Other: Questionnaires — Participants will complete questionnaires to assess activity related dyspnea, respiratory symptoms and health status impairment and respiratory related quality of life.

SUMMARY:
This is a longitudinal study of the long-term impact of COVID-19 on the lungs. Participants will be followed over a period of up to 4 years and impacts of COVID-19 on the lungs will be measured with magnetic resonance imaging (MRI) using hyperpolarized xenon-129, pulmonary function tests, exercise capacity, computed tomography imaging and questionnaires.

DETAILED DESCRIPTION:
This is a multisite longitudinal study of the long-term lung health impact of COVID-19 using hyperpolarized xenon-129 (129Xe) magnetic resonance imaging (MRI) over a period of up to 4 years.

In total 200 participants age ≥ 18 and <80 years who experienced a documented case of COVID-19 (documented by positive COVID-19 test and/or clinical history) will be screened and recruited if they meet all inclusion criteria at the 5 participating sites. Participants will be grouped in mild or severe COVID-19 infection (100 in each group) including 50 with symptoms and at least 50 participants who were hospitalized with COVID-19 infection, all of whom are within 3 months post recovery and non-infectious. Participants will attend up to 5 study visits over the 4 year period. (Visit 1 within 3 months post-COVID-19 recovery, Visit 2 at 24 ± 4 weeks, Visit 3 at 48 ± 4 weeks, Visit 4 at 78 ± 4 weeks, Visit 5 at 200 ± 16 weeks)

At all visits, participants will complete 129Xe MRI, questionnaires (St. George's Respiratory Questionnaire, COPD Assessment Test, Modified Medical Research Council Dyspnea Scale, Modified Borg Scale Breathlessness and Fatigue Questionnaire, Baseline Dyspnea Index Questionnaire and International Physical Activity Questionnaire), pulmonary function tests (Spirometry, Plethysmography, Forced Oscillation Technique, Fractional Exhaled Nitric Oxide, and Multiple Breath Nitrogen Washout), blood and sputum analysis, exercise testing (six-minute walk test). At Visit 1, participants will also complete computed tomography imaging at University Hospital, London Health Sciences Centre. Visits 2 and 4 have the option of being completed over the phone, in which case only questionnaires will be completed. Visit 5 is an optional 4-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are fluent in English reading, understanding and speaking
* Written informed consent must be directly obtained from legally competent participants before any study-related assessment is performed.
* Male and female participants ≥ 18 years and < 80 years.
* Participant experienced a documented case (documented by positive COVID-19 test and/or clinical history) of mild or severe COVID-19 infection.
* Participants are within 3 months post-recovery.
* 100 participants will have had mild symptoms.
* 100 participants will have had severe symptoms, at least 50 of whom were hospitalized.

Exclusion Criteria:

* Participants meeting contraindications for undergoing an MRI such as participants with MRI-sensitive implants, tattoos with MRI-sensitive dye and severe claustrophobia.
* Participant is, in the opinion of the Investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand written material.
* Participant is unable to perform spirometry or plethysmography maneuvers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who experienced a documented mild or severe COVID-19 infection
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by VDP. | 1 year
  Measured using 129-Xenon MRI ventilation defect percent
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by FEV1. | 1 year
  Measured using forced expiratory volume in one second (FEV1)
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by FVC. | 1 year
  Measured using forced vital capacity (FVC)
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by TLC. | 1 year
  Measured using total lung capacity (TLC)
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by FRC. | 1 year
  Functional residual capacity (FRC)
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by RV. | 1 year
  Measured using residual volume (RV)
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by FOT. | 1 year
  Measured using forced oscillation technique (FOT)
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by LCI. | 1 year
  Measured using lung clearance index (LCI)
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by FeNO. | 1 year
  Measured using Fractional Exhaled Nitric Oxide (FeNO).
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by exercise capacity. | 1 year
  Exercise capacity measured by six-minute walk test
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by baseline dyspnea index questionnaire | 1 year
  Measured using the baseline dyspnea index questionnaire.
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by (mMRC) dyspnea scale questionnaire. | 1 year
  Measured using the modified medical research council (mMRC) dyspnea scale questionnaire.
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by CAT. | 1 year
  Measured using the COPD assessment test (CAT).
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by SGRQ. | 1 year
  Measured using the St. George's respiratory questionnaire (SGRQ).
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by IPAQ. | 1 year
  Measured using the International Physical Activity Questionnaire (IPAQ).
Determine long-term respiratory impairment in COVID-19 survivors who did and did not require hospitalization at one year as measured by eosinophil count. | 1 year
  Measured using blood and sputum eosinophil count.

SECONDARY OUTCOMES:
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by VDP. | within 3 months post COVID-19 infection recovery
  Measured using 129-Xenon MRI ventilation defect percent
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by FEV1. | within 3 months post COVID-19 infection recovery
  Measured using forced expiratory volume in one second (FEV1).
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by FVC. | within 3 months post COVID-19 infection recovery
  Measured using forced vital capacity (FVC)
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by TLC. | within 3 months post COVID-19 infection recovery
  Measured using total lung capacity (TLC)
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by FRC. | within 3 months post COVID-19 infection recovery
  Measured using functional residual capacity (FRC)
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by RV. | within 3 months post COVID-19 infection recovery
  Measured using residual volume (RV)
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by FOT. | within 3 months post COVID-19 infection recovery
  Measured using forced oscillation technique (FOT).
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by LCI. | within 3 months post COVID-19 infection recovery
  Measured using lung clearance index (LCI)
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by FeNO. | within 3 months post COVID-19 infection recovery
  Measured using Fractional Exhaled Nitric Oxide (FeNO)
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by exercise capacity. | within 3 months post COVID-19 infection recovery
  Exercise capacity measured by six-minute walk test
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by the baseline dyspnea index questionnaire. | within 3 months post COVID-19 infection recovery
  Measured using the baseline dyspnea index questionnaire.
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by the mMRC dyspnea scale questionnaire. | within 3 months post COVID-19 infection recovery
  Measured using the modified medical research council (mMRC) dyspnea scale questionnaire
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by CAT. | within 3 months post COVID-19 infection recovery
  Measured using the COPD assessment test (CAT)
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by SGRQ. | within 3 months post COVID-19 infection recovery
  Measured using the St. George's respiratory questionnaire (SGRQ)
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by IPAQ. | within 3 months post COVID-19 infection recovery
  Measured using the International Physical Activity Questionnaire (IPAQ).
Determine the clinical, structural, physiologic, and imaging biomarkers within 3 months post COVID-19 infection recovery as measured by eosinophil count.. | within 3 months post COVID-19 infection recovery
  Measured using blood and sputum eosinophil count.
Determine if COVID-19-induced respiratory impairment and predictors of respiratory impairment differ by sex. | up to 4 years
  Evaluated by assessing different genders.
Determine if COVID-19-induced respiratory impairment and predictors of respiratory impairment differ by age. | up to 4 years
  Evaluated by assessing different age groups.
Determine if COVID-19-induced respiratory impairment and predictors of respiratory impairment differ by smoking history measured in pack-years. | up to 4 years
  Evaluated by assessing smoking history measured in pack-years.

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario
Locations (1):
- Department of Medicine (Respirology), McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Health Foundation Workshop on Alcohol and Breast Cancer. December 1, 1987. Proceedings. Prev Med. 1988 Nov;17(6):667-99. No abstract available. PMID 3244666
- [Background] Shukla Y, Wheatley A, Kirby M, Svenningsen S, Farag A, Santyr GE, Paterson NA, McCormack DG, Parraga G. Hyperpolarized 129Xe magnetic resonance imaging: tolerability in healthy volunteers and subjects with pulmonary disease. Acad Radiol. 2012 Aug;19(8):941-51. doi: 10.1016/j.acra.2012.03.018. Epub 2012 May 15. PMID 22591724
- [Background] Schmidt MH, Marshall J, Downie J, Hadskis MR. Pediatric magnetic resonance research and the minimal-risk standard. IRB. 2011 Sep-Oct;33(5):1-6. No abstract available. PMID 22043743
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Oostveen E, MacLeod D, Lorino H, Farre R, Hantos Z, Desager K, Marchal F; ERS Task Force on Respiratory Impedance Measurements. The forced oscillation technique in clinical practice: methodology, recommendations and future developments. Eur Respir J. 2003 Dec;22(6):1026-41. doi: 10.1183/09031936.03.00089403. PMID 14680096
- [Background] Kirby M, Heydarian M, Svenningsen S, Wheatley A, McCormack DG, Etemad-Rezai R, Parraga G. Hyperpolarized 3He magnetic resonance functional imaging semiautomated segmentation. Acad Radiol. 2012 Feb;19(2):141-52. doi: 10.1016/j.acra.2011.10.007. Epub 2011 Nov 21. PMID 22104288
- [Background] Owrangi AM, Etemad-Rezai R, McCormack DG, Cunningham IA, Parraga G. Computed tomography density histogram analysis to evaluate pulmonary emphysema in ex-smokers. Acad Radiol. 2013 May;20(5):537-45. doi: 10.1016/j.acra.2012.11.010. PMID 23570935
- [Background] Pizzichini E, Pizzichini MM, Efthimiadis A, Evans S, Morris MM, Squillace D, Gleich GJ, Dolovich J, Hargreave FE. Indices of airway inflammation in induced sputum: reproducibility and validity of cell and fluid-phase measurements. Am J Respir Crit Care Med. 1996 Aug;154(2 Pt 1):308-17. doi: 10.1164/ajrccm.154.2.8756799.
- [Background] McGavin CR, Artvinli M, Naoe H, McHardy GJ. Dyspnoea, disability, and distance walked: comparison of estimates of exercise performance in respiratory disease. Br Med J. 1978 Jul 22;2(6132):241-3. doi: 10.1136/bmj.2.6132.241. PMID 678885
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Jones PW, Quirk FH, Baveystock CM, Littlejohns P. A self-complete measure of health status for chronic airflow limitation. The St. George's Respiratory Questionnaire. Am Rev Respir Dis. 1992 Jun;145(6):1321-7. doi: 10.1164/ajrccm/145.6.1321. PMID 1595997
- [Derived] Matheson AM, McIntosh MJ, Kooner HK, Abdelrazek M, Albert MS, Dhaliwal I, Nicholson JM, Ouriadov A, Svenningsen S, Parraga G. Longitudinal follow-up of postacute COVID-19 syndrome: DLCO, quality-of-life and MRI pulmonary gas-exchange abnormalities. Thorax. 2023 Apr;78(4):418-421. doi: 10.1136/thorax-2022-219378. Epub 2023 Jan 3. PMID 36596692
- [Derived] Matheson AM, McIntosh MJ, Kooner HK, Lee J, Desaigoudar V, Bier E, Driehuys B, Svenningsen S, Santyr GE, Kirby M, Albert MS, Shepelytskyi Y, Grynko V, Ouriadov A, Abdelrazek M, Dhaliwal I, Nicholson JM, Parraga G. Persistent 129Xe MRI Pulmonary and CT Vascular Abnormalities in Symptomatic Individuals with Post-acute COVID-19 Syndrome. Radiology. 2022 Nov;305(2):466-476. doi: 10.1148/radiol.220492. Epub 2022 Jun 28. PMID 35762891